CLINICAL TRIAL: NCT05077345
Title: The Effects of Different Procedures on Pain Levels at Preterm and Term Infants in Neonatal Intensive Care Unit
Acronym: PAIN
Status: Completed | Type: Observational
Sponsor: Sanko University (Other)
Collaborators: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Hatice Adiguzel, PT, Assistant Proffessor, Kahramanmaras Sutcu Imam University
Other Study IDs: KSU
Record Dates: First submitted 2021-08-16; First posted 2021-10-14 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Pain; Newborn; Preterm; Term; Venipuncture
Keywords: Newborn; pain; Preterm; Term; NICU
MeSH Terms: conditions — Pain; Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- 1/Venous blood sampling: The vessel was determined for cannulation and an anatomical tourniquet was applied. Skin antiseptic was prepared. The plastic wings of the winged angioket were held open. The skin over the vein to be accessed was stretched with the fingers of the free hand. The needle was inserted into the skin a few millimeters distal to the point to be inserted, and the blood was vascularized until the education. The cannula was advanced by retracting the stylet. The tourniquet was removed and the cannula was fixed.
- 2/Heel puncture: The skin was prepared with an antiseptic. The baby's heel was placed at an angle between the thumb and forefinger, with the other fingers grasping the ankle from behind. Pressure was applied to the back of the ankle with the other fingers by taking support against the thumb. The first drop of blood was wiped with sterile gauze by inserting the needle, and the next drops of blood were absorbed into the paper by touching the middle of the ring on the filter paper. An adhesive bandage was applied by applying pressure to the puncture site.
- 3:Orogastric Catheter insertion: The head of the bed was raised and the newborn was placed on his back. The midpoint distance from the tip of the nose to the ear, xiphoid and umbilicus was measured to determine the insertion length. With one hand, the infant's mouth was opened while his head was stabilized. With the other hand, the MV probe was advanced to the specified depth. The position of the OG probe was confirmed and fixed.
- 4:Umbilical Catheter insertion: The system was filled with liquid by connecting the tap to the UK. The faucet was turned off, sterile gauze was placed around the umbilical clamp and lifted out of the sterile area. The other assistant held the cord with a clamp and lifted it vertically up and away from the sterile field. The cord and its surroundings were prepared with an antiseptic solution and covered. The umbilicus was tied with a single knot and the cord was cut horizontally with a scalpel. Bleeding on the surface of the cord was wiped with sterile gauze. The cord stump was grasped with toothed forceps close to the vessel to be catheterized. The catheter was placed in the lumen of the vessel and advanced in the vessel. When the catheter exceeded 5 cm, it was aspirated to confirm the intraluminal position. The blood that came with an average of 0.5 ml bolus solution was cleaned and the catheter was fixed.
- 5:Tracheal Intubation: The head of the infant was positioned in the midline, slightly extended, with the chin up. The head was stabilized with the right hand by turning on the light of the laryngoscope. The blade of the laryngoscope was inserted by sliding the blade over the tongue until the tip of the blade rested on the Vallecula. The blade of the laryngoscope was slid up to open the mouth even more. The other assistant gently dipped it into the suprasternal notch. The concave edge of the tube was held with the right hand, and it was advanced approximately 2 cm, passing it between the vocal cords when the vocal cords and trachea were seen.

SUMMARY:
Accurate assessment of pain in neonates in the neonatal intensive care unit (NICU) is vital because of the high prevalence of painful experiences, including both daily procedural pain and postoperative pain, in this population. It has been reported that newborns born between the gestational ages (GY) 25-42 and hospitalized in the NICU undergo an average of 14 painful procedures per day in the first 2 weeks of life. The aim of this study is determinin the effect of different procedures on the pain levels of newborns in the Neonatal Intensive Care Unit (NICU).

DETAILED DESCRIPTION:
Accurate assessment of pain in neonates in the neonatal intensive care unit (NICU) is vital because of the high prevalence of painful experiences, including both daily procedural pain and postoperative pain, in this population. Exposure of these infants to many mandatory invasive procedures and poor pain management during this time may lead to different results in the short and long term. Every painful application in newborns causes behavioral and physiological instability. Repeated exposure to painful stimuli produces long-term changes in stress-sensitive brain systems such as the hypothalamic-adrenal system and the developing brain. Therefore, evaluation and prevention of pain in newborns is essential. In the NICU, many medical interventions are often performed on infants that are repetitive, painful, but diagnostically necessary. All environmental stress factors can cause physiological changes such as increased pulse, blood pressure, respiratory rate and a decrease in oxygen saturation in newborns. Increasing energy expenditure to overcome these changes may affect physiological functioning, slowing recovery and adversely affecting the organization of the central nervous system (CNS). Heel blood (TC), vascular access (DY), naso and orogastric (NG-OG) catheter insertion, arterial blood collection, tracheal intubation (TE), various rectal procedures, removal of adhesive tapes, umbilical catheter (UK) insertion and removal, Various procedures such as aspiration, chest physiotherapy applications, diaper changing, various hand contacts, and general body care may induce pain responses in newborns. While these responses are associated with low cognitive and motor scores in early childhood, they may result in changes in visual-perceptual ability and somatosensory sensitivity later on. There are many studies in the literature to increase and prove the accuracy of pain assessment tools. However, since the pain treatments used in these studies were also varied, the homogeneity of the evaluations was insufficient. Therefore, more systematic evaluation studies should be conducted on how to improve pain management in NICUs. Finding which of the painful stimuli affects infants more will also guide the use of treatment methods. The aim of this study is to investigate the effects of different procedures applied in the NICU on the pain levels of term and preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* Preterm and term infants admitted to the NICU for the first time for various reasons with a hospital stay ranging from 1 to 8 days
* Preterm and term infants who were cared for in an incubator without any pharmacological or non-pharmacological analgesic therapy, muscle relaxant, and sedation treatment in the last 24 hours before the procedure.

Exclusion Criteria:

* Exposed to painful procedures more than 3 times in the same day
* Infants who diagnosed with osteomyelitis, sepsis, pyejonic arthritis, congenital anomaly (Spina bifida, arthrogryposis multiplex congenita)
* Infants with any known neurological diagnosis (Abnormal MRI finding, hydrocephalus, Chiari malformation, asphyxia, periventricular leukomolacia (PVL), acute bilirubin encephalopathy, hypoxic ischemic encephalopathy (HIE))
* Infants who had any surgery

Ages: 1 Day to 8 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study included 196 newborns who were hospitalized in SANKO University Hospital Level 3 NICU and exposed to different painful procedures during routine clinical practices under Neonatologist follow-up.
Sampling Method: Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Neonatal Infant Pain Scale | The pain scale was scored in the first 5 minutes following the clinical procedure.
  pain measurement of infants. This scale measures five behavioral groupings (i.e. facial expressions, crying, movements of arms and legs, and awake condition), and one physiological parameter (i.e. breathing patterns) given against pain during invasive procedures in preterm and term infants. The total score is between "0" and "7". The lowest pain level is 0, and the highest pain level is 7. The validity and reliability of the scale were shown in studies that were conducted with premature and term newborns.
O₂ saturation1 | O₂ saturation value of the newborn 5 minutes before the painful procedure from the pulse oximeter.
  O₂ saturation of the newborn 5 minutes before the painful procedure.
heart rate1 | the heart rate of the newborn 5 minutes before the painful procedure from the monitor
  the heart rate of the newborn 5 minutes before the painful procedure
heart rate2 | the heart rate of the newborn at the time point of the painful procedure from the monitor
  the heart rate of the newborn during the painful procedure
heart rate3 | the heart rate of the newborn 5 minutes after the painful procedure from the monitor
  the heart rate of the newborn 5 minutes after the painful procedure
O₂ saturation2 | O₂ saturation of the newborn at the time point of the painful procedure from the pulse oximeter.
  O₂ saturation of the newborn during the painful procedure.
O₂ saturation3 | O₂ saturation of the newborn 5 minutes after the painful procedure from the pulse oximeter.
  O₂ saturation of the newborn 5 minutes after the painful procedure.

SECONDARY OUTCOMES:
The type and Number of painful procedures | The type and number of painful procedures during the first 8 days of life performed on newborns were also recorded.
  The type and number of painful procedures will be recorded as Heel Puncture (HP), Venous Blood sampling (VB), naso and orogastric (NG-OG) catheter insertion, arterial blood collection, Tracheal Intubation (TI), several rectal procedures, the removal of adhesive tapes, insertion and removal of Umbilical Catheter (UC), and several other procedures such as aspiration, chest physiotherapy procedures,
age (day) | up to 7 days
  age of the infants will be recorded as day.
length (centimeter/cm) | It will be recorded on the pain assesment day.
  birth length of the infants
gender | up to 7 days
  gender of the infants will be recorde as f/m
Diagnosis of the infants (the reason for hospitalization of the infants) | up to 7 days
  the reason for hospitalization of the infants will be recorded as Prematurity, Respiratuar Distress Syndrome (RDS), Bronchopulmonary Dysplasia (BPD), Low birth weight (LBW), Extreme low birth weight (ELBW), Sepsis, Patent Ductus Arteriosus (PDA), Retinopathy of Prematurity (ROP), Small for gestational age (SGA), Premature Rupture of Membranes (PROM).
the duration (day) of hospitalization of infants | up to 7 days
  the duration of hospitalization of all infants will be recorded as day.
birth weight | at birth
  birth weight will be recorded in kilograms(kg)

CONTACTS AND LOCATIONS:
Overall Officials: hatice Adiguzel, PhD, Principal Investigator — Kahramanmaras Sutcu Imam University; mehmet Egilmez, PT, Study Chair — Sanko University; Nevin Ergun, Proffessor, Study Chair — Sanko University; Yusuf Unal Sarıkabadayi, Doctor, Study Chair — Sanko University; Bulent Elbasan, Proffessor, Study Director — Gazi University
Locations (1):
- Hatice Adıgüzel, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No